CLINICAL TRIAL: NCT06673004
Title: Ovarian Tissue Allo-Transplantation in the Setting of Primary Ovarian Insufficiency Between Non-Genetically Identical Siblings With Use of Immunosuppression
Brief Title: Ovarian Tissue Allo-transplantation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecca Flyckt (Other)
Responsible Party: Sponsor-Investigator, Rebecca Flyckt, Division Chief, Reproductive Endocrinology and Infertility, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20241094
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Failure; Ovarian Insufficiency; Menopause Ovarian Failure; Menopause, Premature; Infertility, Female; Endocrine Female Infertility
Keywords: Primary ovarian insufficiency; Ovarian tissue transplantation; Immunosuppression; Premature menopause; Ovarian failure; Ovary transplant
MeSH Terms: conditions — Menopause, Premature; Infertility, Female; Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ovarian tissue recipient (Experimental): Any recipient that receives ovarian tissue transplantation
  Interventions: Procedure: Ovarian tissue allo-transplantation

INTERVENTIONS:
Procedure: Ovarian tissue allo-transplantation — Participants will receive donor ovarian tissue with immunosuppression

SUMMARY:
Premature ovarian failure, also known as primary ovarian insufficiency (POI), or premature menopause, affects 1-2% of women under 40. The diagnosis is typically made based on high levels of follicle stimulating hormone (FSH) and absent or irregular menstrual periods. It leads to infertility and menopause-like effects (hot flashes and thin bones) due to low estrogen levels. POI can result from various factors such as genetic conditions, autoimmune diseases, or previous medical treatments like chemotherapy.

Treatment of POI usually involves hormone replacement therapy and, if pregnancy is desired, assisted reproductive technologies such as in vitro fertilization (IVF) using an egg donor. However, IVF may not be an option for everyone due to personal, religious, ethical or financial reasons. Recent advances in medicine have identified ovarian tissue transplantation (OTT) as a potential solution. OTT involves transplanting either fresh or frozen ovarian tissue into the pelvic area, where it can begin functioning again. Studies in animals and humans have shown success in restoring hormonal function and even achieving pregnancies in some cases. Initial human trials of ovarian tissue transplants from another individual began with identical twins and have since expanded to include non-identical siblings with compatible tissue matches using immunosuppression. Success rates of OTT have been promising, with multiple live births reported between identical twins. Long-term studies indicate that transplanted tissue can remain functional for up to eight years. Ovarian tissue transplantation offers a promising avenue for women with POI to help restore fertility and hormonal function. Continued research and refinement of tissue techniques are essential to improve outcomes and expand access to this innovative treatment option.

This study will enroll 10 participants who will undergo ovarian tissue transplantation donated by a non-identical sister using an immunosuppression protocol at University Hospitals.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Must meet criteria for primary ovarian insufficiency
* Amenorrheic x12 months
* Serum hormone (FSH, LH, estradiol, AMH) levels consistent with menopause
* Must be between the ages of 21-40 years old.
* Must be in a committed relationship with a male partner.
* Must be willing to attempt natural conception within 4 months following transplant.
* Must be willing to undergo a pre-transplant evaluation.
* Must be willing to undergo Maternal Fetal Medicine consultation and evaluation for safety of pregnancy, particularly patients at risk of complications in pregnancy (e.g. Turner syndrome patients).
* Must be willing to undergo general anesthesia, minimally invasive gynecologic surgery, pregnancy with potential high risk complications, and surgery to remove the graft
* Must be willing and able to receive potent immunosuppressive medications and must be able to follow standard infection prophylaxis protocols
* Must be willing to receive standard vaccinations such as influenza, Hepatitis B. If age and circumstances indicate, be willing to receive vaccines against pneumococcus, HPV and Hepatitis A.
* If patient is a smoker, 3 months cessation is required prior to enrollment and must pass a nicotine test.
* Must be willing and able to sign informed consent and follow all outlined procedures and recommendations in the protocol, including assent for monitoring neonatal outcomes for the first year after birth.

Recipient Exclusion Criteria:

* History of hypertension, diabetes, or significant heart, liver, kidney or central nervous system disease. Serum creatinine level >1.0 mg/dL.
* Any medical diagnosis placing the subject at high risk of surgical complications based on the team's review of medical history.
* Current smoker (smoking cessation must have occurred 3 months prior to enrollment).
* Active HPV infection.
* History of prior malignancy except for cervical cancer in stage 1a or 1b after 3 years.
* History of human immunodeficiency virus (HIV), mycobacteria, hepatitis C.
* Hepatitis B infection (Hepatitis B risk is for those with HepB surface antigen and/or HBV DNA positive. Those that are HepB core antibody true-positive are at minimal risk of reactivation. Those with vaccine-induced HepB surface antibody are not at risk).
* Presence of active documented systemic infection or recent systemic infection within the past three months.
* Chemical and/or alcohol dependency or abuse.
* BMI greater than 30 kg/m2
* Prior organ transplant with rejection, infection, or graft thrombosis.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-05-30 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Time (days) from transplantation to resumption of menses as measured by patient report | Up to 6 months
Number of live births as measured by medical record report/patient report | Up to 3 years

SECONDARY OUTCOMES:
Time (days) from transplantation to pregnancy as measured by medical record/patient report | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Flyckt, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Kathryn Coyne, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No